CLINICAL TRIAL: NCT05576467
Title: Treatment for Migraine and Mood (TEAM-M): A Randomized Controlled Trial of a Mindfulness-based Training Program
Brief Title: Treatment for Migraine and Mood
Acronym: TEAM-M
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amanda Shallcross (Other)
Collaborators: Yeshiva University (Other); Wake Forest University Health Sciences (Other); The Cleveland Clinic (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Amanda Shallcross, Associate Professor of Medicine, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20225608; R01AT011005 (NIH)
Record Dates: First submitted 2022-10-10; First posted 2022-10-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-06

CONDITIONS: Migraine; Depressive Symptoms
Keywords: mindfulness; mindfulness-based cognitive therapy
MeSH Terms: conditions — Migraine Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MBCT-Telephone (Active Comparator): 8 weekly classes delivered via telephone.
  Interventions: Behavioral: MBCT-Telephone
- MBCT-Video (Active Comparator): 8 weekly classes delivered via video.
  Interventions: Behavioral: MBCT-Video
- Enhanced Usual Care (EUC) (Active Comparator): 8 weekly online modules delivered via web portal.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: MBCT-Telephone — Classes follow MBCT protocol delivered via telephone by a master's level or higher mental health provider under the supervision of a licensed clinical psychologist, following treatment fidelity guidelines from NIH's Behavioral Change Consortium.
  Arms: MBCT-Telephone
Behavioral: MBCT-Video — Classes follow MBCT protocol delivered via video by a master's level or higher mental health provider under the supervision of a licensed clinical psychologist, following treatment fidelity guidelines from NIH's Behavioral Change Consortium.
  Arms: MBCT-Video
Behavioral: Enhanced Usual Care (EUC) — Weekly online modules follow migraine and behavior principles delivered via web portal developed by a team of licensed clinical psychologists, neurologists, and mental health providers.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The researchers propose a three-arm pilot study of Mindfulness-Based Cognitive Therapy (MBCT) delivered via telephone (MBCT-T), video (MBCT-V) or Enhanced Usual Care (EUC).

DETAILED DESCRIPTION:
This study aims to set the stage for a future definitive large-scale Phase III trial in patients with migraine and depressive symptoms. This pilot is aimed at evaluating the feasibility and acceptability of the Telephone and Video MBCT and EUC in people with migraine (defined by the International Classification of Headache Disorders - 3) and depressive symptoms (defined by empirical cut-offs on the Patient Health Questionnaire - 9).

ELIGIBILITY:
Inclusion Criteria:

* Currently meets ICHD-3 (International Classification for Headache Disorders - 3rd Edition) criteria for migraine using the American Migraine Prevalence and Prevention Diagnostic Module
* Self-reported 4-14 headache days per month, with at least one attack meeting migraine criteria
* Score between 5-14 on the PHQ-9 (Patient Health Questionnaire)
* Age ≥ 18
* Ability to read and speak English
* Capacity to consent
* Prospective diary-confirmed 4-14 headache days per month, with at least one attack meeting migraine criteria
* ≥1 year of migraine

Exclusion Criteria:

* Meeting ICHD-3 criteria for persistent headache attributed to traumatic injury to the head (post-traumatic headache) on the American Migraine Prevalence and Prevention Diagnostic Module
* Changes in preventive migraine medication or anti-depressant medication within 6 weeks of intake
* Changes in longer-term migraine prevention (onabotulinum toxin A, injectable or oral anti-calcitonin gene related peptide treatment; neuromodulatory device) within 3 months of intake
* Changes in acute migraine treatment started within 4 weeks of enrollment
* Comorbid psychiatric illness or clinical features that would interfere with participant's ability to participate in or receive benefit from the intervention, including but not limited to: active suicidal ideation; recent history of psychosis or mania; borderline, histrionic or narcissistic personality disorder; cognitive impairment; sensory disabilities; bipolar disorder; obsessive-compulsive disorder, drug use
* Prior history of engaging in formal mindfulness-based interventions including: MBSR (Mindfulness-based stress reduction), MBCT (Mindfulness-based cognitive therapy), Acceptance and Commitment therapy, Dialectical Behavior Therapy
* Current daily meditation practice
* Inability to adhere to headache diary during baseline evaluation period (recorded fewer than 25/28 days)
* Unwilling to maintain stable current acute or preventive medication dosages for study duration
* Any condition that would prevent being a suitable candidate or interfere with medical care needs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2024-03-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of Treatment Session Adherence | Week 8
  Treatment Session Adherence is a measure of treatment feasibility. This measure will be assessed through electronic monitoring of the attendance logs of each treatment session. The number of treatment sessions attended will be recorded. A treatment arm will be considered feasible if participants attended/read 75% of sessions on average.
Client Satisfaction Questionnaire - 8 (CSQ-8) | Week 8
  The CSQ-8 assesses treatment acceptability. The CSQ-8 is an 8-item self-report measure designed to assess satisfaction with mental health services. Response options are coded on a 4-point scale and summed to produce a total score ranging from 8-32. The measure has consistently demonstrated excellent reliability and validity, and is commonly used in behavioral treatment trials. For the purposes of this study, a CSQ-8 score > 24 is considered acceptable.

SECONDARY OUTCOMES:
Change in Headache Disability Inventory (HDI) | Month 0 to Month 3
  The HDI is a 25-item self-report survey which assesses perceived emotional and functional impact of headache on daily activities. Sample items include, "Because of my headaches I feel restricted in performing my routine daily activities," with response options of "Yes," "Sometimes," and "No." Total scores range from 0-100, with higher scores indicating higher disability. The slope of change between Month 0 and 3 represents a secondary outcome designed to evaluate clinical signal in this pilot study.
Change in Migraine-Specific Quality of Life Questionnaire v 2.1 (MSQ) | Month 0 to Month 3
  The MSQ is a 14-item self-report survey which assesses quality of life over the past 4 weeks in people with migraine. Items comprise three subscales: Role Restriction, Role Prevention, and Emotion Function. Each item is scored on a Likert-type scale from 1 ("None of the time") to 6 ("All of the time"). Total scores range from 14-84. The slope of change between Month 0 and 3 represents a secondary outcome designed to evaluate clinical signal in this pilot study.
Change in Quick Inventory of Depressive Symptomatology - Self-Report 16 (QIDS-SR16) | Month 0 to Month 3
  The QIDS-SR16 measures depressive symptom domains during the prior 7 days. Each item is scored on a scale from 0 to 3 points. Total scores range from 0 to 27. Score cutoffs are: 1-5 for no depression, 6-10 for mild depression, 11-15 for moderate depression, 16-20 for severe depression, and 17-27 for very severe depression. The slope of change between Month 0 and 3 represents a secondary outcome designed to evaluate clinical signal in this pilot study.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Seng, Ph.D., Principal Investigator — Albert Einstein College of Medicine and Yeshiva University; Amanda J Shallcross, M.P.H., N.D., Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - Albert Einstein College of Medicine, The Bronx, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available upon request to qualified individuals in the research community. If this research develops or improves any technologies or techniques, this work will be made available to qualified individuals in the research community.
Supporting Information: Study Protocol
Time Frame: Individual participant data will become available at the conclusion of the study upon request by qualified individuals in the research community.